CLINICAL TRIAL: NCT02355327
Title: Feasibility Trial on the Effectiveness of Vibrating Vaginal Balls to Improve Pelvic Floor Muscle Performance in Women After Childbirth
Brief Title: Vibrating Vaginal Balls After Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SREC 14-15 02 D 02 12 2014; 1704/2014 (Other: Medical University of Vienna)
Record Dates: First submitted 2015-01-13; First posted 2015-02-04 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-01

CONDITIONS: Pelvic Floor Health After Childbirth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laselle Kegel Exerciser (Experimental)
  Interventions: Device: Laselle Kegel Exerciser
- Pelvic floor muscle exercises (Active Comparator)
  Interventions: Behavioral: Pelvic floor muscle exercises

INTERVENTIONS:
Device: Laselle Kegel Exerciser — Participants use a vibrating pelvic floor muscle training ball for 12 weeks. The ball is inserted into the vagina and left for 15 minutes daily in the first week, and if well tolerated 30 minutes daily from the second week onwards. To achieve the vibrating effect, the balls are worn while moving - performing everyday tasks or going for a walk.
  Arms: Laselle Kegel Exerciser
Behavioral: Pelvic floor muscle exercises — Participants get standard care after childbirth, which is the routine recommendation of pelvic floor muscle exercises. Participants will be asked to continue/start the pelvic floor muscle exercises they routinely were recommended by customary written instructions from their health professionals after birth. Intervention duration for this study is 12 weeks.
  Arms: Pelvic floor muscle exercises

SUMMARY:
This feasibility trial aims at assessing practical issues and feasibility of a future randomised controlled trial (RCT) to determine the effectiveness of vibrating vaginal pelvic floor training balls for postpartum pelvic floor muscle rehabilitation, at monitoring harms of the experimental intervention, and at exploring women´s perspectives on and experiences with the interventions and the trial.

DETAILED DESCRIPTION:
Background: Pelvic floor muscle training after childbirth is recommended to prevent or treat urinary incontinence and other pelvic floor problems. A device that is sometimes recommended to women in Austria to enhance their pelvic floor muscles are vibrating vaginal pelvic floor training balls. To date, only a small study on vibrating balls exists, and it researched women with urinary incontinence and not women after childbirth. Therefore, research is needed to scientifically objectify the popular claim of these balls´ effectiveness in the postpartum period and further evidence based practice.

Method: The tested study features comprise

* recruitment strategies,
* inclusion and exclusion criteria,
* the necessary number of participants,
* the randomisation procedure,
* the interventions themselves,
* concordance and retention measures,
* data collection,
* effectiveness outcomes,
* a survey of women's views of and experiences,
* statistics and content analysis.

Results: The results of this trial will inform the features and feasibility of a future full RCT. It will be concluded that a full RCT to determine the effectiveness of vibrating vaginal pelvic floor training balls post partum is feasible as planned, feasible with modifications or not feasible. If considered feasible, the results will enable the full study to be planned correctly.

ELIGIBILITY:
Inclusion Criteria:

* Women from 6 weeks to 6 months after vaginal childbirth (at beginning of intervention)
* Term birth, i.e. 37+0 or more weeks of gestation
* 6 weeks postpartum check by obstetrician-gynaecologist performed and woman discharged from postpartum care with diagnostic findings appropriate to this period after childbirth
* Lochia have ceased
* Baby alive/not seriously ill
* Sufficient knowledge of written and spoken German to be able to participate in the study
* Capacity to consent

Exclusion Criteria:

* Currently enrolled in pelvic floor muscle training with physiotherapist, midwife or fitness trainer
* Status post perineal tear 3rd or 4th degree at most recent birth
* Status post continence surgery
* Current pelvic floor or gynaecological surgery
* Current infection of genitourinary tract
* Recurrent (>5 infectious episodes during last 12 months) or chronic (>3 weeks duration of single episode in last 12 months) vaginal infections
* Neuromuscular conditions influencing pelvic floor muscle function (e.g. multiple sclerosis)
* Major medical condition influencing infectious risk (diabetes, immune suppressive therapy, HIV infection etc.)
* Currently on medication that could interfere with treatment or evaluation
* Currently enrolled in any other research study
* Pregnancy (also commencing during participation) or pregnancy planned within the study period
* Retention of ball is impossible
* Inability to perform the proposed procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by recruitment rate | Within 4 weeks of ending recruitment
Feasibility as measured by pre intervention pelvic floor muscle measurement attendance rate | Within 4 weeks of ending data collection
Feasibility as measured by start of intervention rate | Within 4 weeks of ending data collection
Feasibility as measured by concordance rate | Within 4 weeks of ending data collection
Feasibility as measured by retention rate | Within 4 weeks of ending data collection
Feasibility as measured by post intervention data collection attendance rate | Within 4 weeks of ending data collection
Feasibility as measured by staff necessary | Within 4 weeks of ending data collection
Feasibility as measured by time necessary | Within 4 weeks of ending data collection
Feasibility as measured by budget necessary | Within 4 weeks of ending data collection

OTHER OUTCOMES:
Participant reported pelvic floor muscle outcomes as measured by structured questionnaire | Within 3 weeks before the intervention
  Questionnaire contains self-designed section and also includes the International Consultation on Incontinence Modular Questionnaire Urinary Incontinence Short Form (ICIQ UI)
Participant reported pelvic floor muscle outcomes as measured by structured questionnaire | Within 2 weeks after the intervention
  Questionnaire contains self-designed section and also includes the International Consultation on Incontinence Modular Questionnaire Urinary Incontinence Short Form (ICIQ UI)
Pelvic floor muscle performance as measured by perineometry | Within 4 days before the intervention
  By blinded external assessor
Pelvic floor muscle performance as measured by perineometry | Within 2 weeks after the intervention
  By blinded external assessor
Women´s perspectives and experiences as measured by structured interviews | Within 3 weeks before the intervention
  28 of 56 women
Women´s perspectives and experiences as measured by structured interviews | Within 2 weeks after the intervention
  Same 28 of 56 women as for previous outcome measure
Women´s perspectives and experiences as measured by structured anonymous questionnaire | Within 3 weeks after the intervention
  28 of 56 women (those not included in the two previous outcome measures)
Concordance to interventions as measured by training diary | At time of intervention (12 weeks)
Type, severity and number of adverse events as measured by active and passive surveillance (interview, self-report) | At time of intervention (12 weeks)
Type, severity and number of adverse events as measured by active and passive surveillance (interview/questionnaire, self-report) | Up to 1 year after end of intervention
  First 28 of 56 women: interview, second 28 of 56 women: questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Oblasser, MA, cand.PhD, Principal Investigator — City, University of London; Engelbert Hanzal, MD, Prof., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Oblasser C, Christie J, McCourt C. Vaginal cones or balls to improve pelvic floor muscle performance and urinary continence in women postpartum: a quantitative systematic review and meta-analysis protocol. J Adv Nurs. 2015 Apr;71(4):933-41. doi: 10.1111/jan.12566. Epub 2014 Nov 10. PMID 25382375
- [Background] Oblasser C, Christie J, McCourt C. Vaginal cones or balls to improve pelvic floor muscle performance and urinary continence in women post partum: A quantitative systematic review. Midwifery. 2015 Nov;31(11):1017-25. doi: 10.1016/j.midw.2015.08.011. Epub 2015 Sep 9. PMID 26428191
- [Background] Oblasser C, McCourt C, Hanzal E, Christie J. Vibrating vaginal balls to improve pelvic floor muscle performance in women after childbirth: a protocol for a randomised controlled feasibility trial. J Adv Nurs. 2016 Apr;72(4):900-14. doi: 10.1111/jan.12868. Epub 2015 Dec 28. PMID 26708615
- See also: Entry at study registry of the Ethics Committee of the Medical University of Vienna — https://ekmeduniwien.at/core/catalog/2014/